CLINICAL TRIAL: NCT01123668
Title: Neuropharmacology of Response Inhibition in Comorbid ADHD and Nicotine Dependence
Brief Title: Neuroimaging of Smokers With and Without Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00009085; 1R01DA024838-01A1 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2014-08

CONDITIONS: Smoking; ADHD
Keywords: Smoking; ADHD; Nicotine; Methylphenidate; function Magnetic Resonance Imaging; Neurobiological basis of abstinence-induced deficits in response inhibition
MeSH Terms: conditions — Smoking; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples With DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADHD and non-ADHD Smokers: Those that are defined as regular smokers (10 cigarettes/day or Carbon Monoxide reading of 10 ppm). The group will then be split into those diagnosed with ADHD/ADD and controls for comparison.

SUMMARY:
The purpose of this study is to evaluate how nicotine, withdrawal from nicotine, and methylphenidate (a drug used for the treatment of ADHD) affect the brain of smokers with and without ADHD while doing tasks in an functional Magnetic Resonance Imaging scanner.

Study Hypotheses:

1. compared to non-ADHD smokers, smokers with ADHD will exhibit greater abstinence-induced decrements in response inhibition performance and reward and greater concomitant disruptions of brain activity
2. administration of MPH to abstinent smokers will ameliorate response inhibition performance and reward deficits and task-related brain activation and this effect will be greater among ADHD smokers
3. genetic markers of dopamine neurotransmission will moderate abstinence- and MPH - induced changes in task-related brain activation across tasks.

DETAILED DESCRIPTION:
Individuals diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) smoke more than the general population, initiate use at a younger age, and report more difficulty trying to quit. The overarching goal of the present application is to use neuroimaging, neuropharmacological and molecular genetic techniques to study the neurobiological basis of abstinence-induced deficits in response inhibition in ADHD and non-ADHD smokers. Twenty smokers with ADHD and 20 smokers without ADHD will undergo imaging during a Go/No-Go task under the following conditions: 1) smoking as usual, 2) 24 hr smoking abstinence, and 3) 24 hr smoking abstinence + methylphenidate (MPH). We hypothesize that compared to smoking as usual, 24 hr smoking abstinence will result in decrements in response inhibition and disruption of task-related brain activation. These effects will be greater in ADHD as compared to non-ADHD smokers. We further hypothesize that MPH administration during abstinence will restore performance and brain indices of response inhibition and that the magnitude of the effect of MPH will be greater among smokers with ADHD. In addition to the above aims, we will preliminarily evaluate the moderating effects of the dopamine receptor D4 7-repeat allele on task-related brain activation following smoking abstinence and MPH administration.

During the study, 101 subjects signed consents and 38 subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. generally healthy, between the ages of 18-50yrs,
2. smoking at least 10 cigarettes/day of a brand delivering ≥0.5 mg nicotine according to the standard Federal Trade Commission (FTC) method,
3. an expired Carbon Monoxide concentration of at least 10ppm (to confirm inhalation) or a positive urine cotinine test (Nicalert ™) of 3 or greater,
4. no interest in quitting smoking as measured by self-report,
5. right-handed as measured by a three item scale used in our laboratory.

Exclusion Criteria:

1. unable to attend all required experimental sessions,
2. have significant health problems (e.g., chronic hypertension, emphysema, seizure disorders, history of significant heart problems),
3. use of psychoactive medications with the exception of ADHD pharmacotherapies among ADHD diagnosed participants (see washout procedures below)
4. use of smokeless tobacco
5. current or past year alcohol or drug abuse,
6. use of illegal drugs as measured by urine drug screen or self report
7. current use of nicotine replacement therapy or other smoking cessation treatment,
8. presence of conditions that would make MRI unsafe (e.g., pacemaker, metal objects in the body, IUD),
9. if they are female and pregnant or plan on becoming pregnant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 120 voluntary participants to yield 40 Adult Regular Smokers, including 20 diagnosed with ADHD and 20 comparison controls.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2009-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of smoking abstinence on response inhibition brain function in smokers with and without ADHD. | July 2009 through December 2013
  Smokers will undergo three functional Magnetic Resonance Image scanning sessions while performing a task that measures response inhibition (Go/Go/No-Go task) Scanning will take place in the following conditions: smoking as usual + placebo pill, 24 hr smoking abstinence + placebo pill and 24 hr abstinence + methylphenidate (MPH). Methylphenidate is a dopamine reuptake inhibitor and its administration will allow us to evaluate the role of dopamine neurotransmission on response inhibition in the context of smoking abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D., Principal Investigator — Duke Health
Locations (1):
- Duke Child and Family Study Center//Duke Health Behavior Neuroscience Research Program, Durham, North Carolina, United States